CLINICAL TRIAL: NCT01629498
Title: Phase I/II Trial of Image-Guided, Intensity-Modulated Photon (IMRT) or Scanning Beam Proton Therapy (IMPT) Both With Simultaneous Integrated Boost (SIB) Dose Escalation to the Gross Tumor Volume (GTV) With Concurrent Chemotherapy for Stage II/III Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Image-Guided, Intensity-Modulated Photon or Proton Beam Radiation Therapy in Treating Patients With Stage II-IIIB Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-1058; NCI-2012-01224 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2011-1058 (Other: M D Anderson Cancer Center); P01CA021239 (NIH); U19CA021239 (NIH)
Record Dates: First submitted 2012-06-25; First posted 2012-06-27 (Estimated); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Lung Non-Small Cell Carcinoma; Stage II Non-Small Cell Lung Cancer AJCC v7; Stage IIA Non-Small Cell Lung Carcinoma AJCC v7; Stage IIB Non-Small Cell Lung Carcinoma AJCC v7; Stage IIIA Non-Small Cell Lung Cancer AJCC v7; Stage IIIB Lung Non-Small Cell Cancer AJCC v7
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy, Image-Guided; Radiotherapy, Intensity-Modulated; Proton Therapy; Protons

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (image-guided IMRT) (Experimental): Patients undergo image-guided IMRT SIB QD 5 days a week for up to 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: Image Guided Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Radiation: Photon Beam Radiation Therapy; Other: Questionnaire Administration
- Arm II (image-guided IMPT) (Experimental): Patients undergo image-guided IMPT SIB QD 5 days a week for up to 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: Image Guided Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Radiation: Proton Beam Radiation Therapy; Other: Questionnaire Administration

INTERVENTIONS:
Radiation: Image Guided Radiation Therapy — Undergo image-guided IMRT
  Other Names: IGRT; image-guided radiation therapy
  Arms: Arm I (image-guided IMRT)
Radiation: Image Guided Radiation Therapy — Undergo image-guided IMPT
  Other Names: IGRT; image-guided radiation therapy
  Arms: Arm II (image-guided IMPT)
Radiation: Intensity-Modulated Radiation Therapy — Undergo image-guided IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy
  Arms: Arm I (image-guided IMRT)
Radiation: Intensity-Modulated Radiation Therapy — Undergo image-guided IMPT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy
  Arms: Arm II (image-guided IMPT)
Other: Laboratory Biomarker Analysis — Optional correlative studies
Radiation: Photon Beam Radiation Therapy — Undergo image-guided IMRT
  Arms: Arm I (image-guided IMRT)
Radiation: Proton Beam Radiation Therapy — Undergo image-guided IMPT
  Other Names: PBRT; Proton Radiation Therapy
  Arms: Arm II (image-guided IMPT)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This partially randomized phase I/II trial studies the side effects and best dose of image-guided, intensity-modulated photon or proton beam radiation therapy and to see how well they work in treating patients with stage II-IIIB non-small cell lung cancer. This trial is testing a new way of delivering radiation dose when only the tumor receives dose escalation while the surrounding normal structure is kept at standard level. Photon beam radiation therapy is a type of radiation therapy that uses x-rays or gamma rays that come from a special machine called a linear accelerator (linac). The radiation dose is delivered at the surface of the body and goes into the tumor and through the body. Proton beam radiation therapy is a type of radiation therapy that uses streams of protons (tiny particles with a positive charge) to kill tumor cells. Both methods are designed to give a higher than standard dose of treatment to the tumor and may reduce the amount of radiation damage to healthy tissue near a tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the maximum tolerated dose (MTD) of image-guided intensity-modulated photon (IMRT) and proton therapy (IMPT) both with simultaneous integrated boost (SIB) dose escalation to the SIBVi (internal SIB volume; defined as the gross tumor volume with consideration of respiratory motion plus setup uncertainty margin) for patients with stage II/IIIB non-small cell lung cancer (NSCLC) receiving concurrent standard chemotherapy and proton irradiation. (Phase I) II. Assess and compare survival free of grade III treatment related toxicity and local progression-free survival from day 1 of concurrent chemoradiation for stage II-IIIB NSCLC patients treated with image-guided robustly-optimized IMPT versus (vs.) IMRT, both delivered with simultaneous integrated boost (SIB). (Phase II)

SECONDARY OBJECTIVES:

I. Determine treatment-related acute and late toxicity. II. Correlate changes in standardized uptake values (SUV) on positron emission tomography (PET) and study endpoints (toxicity, tumor response, local control).

III. Correlate changes in peripheral blood biomarkers (genes, micro-ribonucleic acid [RNA], proteins) and the study endpoints.

IV. Estimate progression-free and overall survival. V. Document and compare symptom burden before starting chemoradiation, weekly during treatment, bi-weekly from end of treatment until first follow up, and at each follow-up visit thereafter by using the MD Anderson Symptom Inventory - Plus (MDASI-Plus) and European Quality of Life Instrument-5 dimensions (EQ-5D).

VI. Perform cost effectiveness between IMPT and IMRT both with SIB treatment. VII. Correlate imaged response, clinical response, blood biomarkers and symptom burdens to dose distribution patterns.

OUTLINE: This is a phase I, dose-escalation study followed by a randomized phase II study.

PHASE I: Patients undergo image-guided IMRT with SIB or IMPT with SIB once daily (QD) 5 days a week for up to 6 weeks in the absence of disease progression or unacceptable toxicity.

PHASE II: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients undergo image-guided IMRT SIB QD 5 days a week for up to 6 weeks in the absence of disease progression or unacceptable toxicity.

ARM II: Patients undergo image-guided IMPT SIB QD 5 days a week for up to 6 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 4-8 weeks, every 3-4 months for 3 years, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven diagnosis of unresected stage II-IIIB, or recurrent after surgical resection or stereotactic body radiation therapy (SBRT) non-small cell lung cancer
* Suitability for concurrent chemoradiation therapy per treating physician's assessment
* Karnofsky performance status (KPS) score >= 70
* Weight loss < 15% in the 3 months before diagnosis
* Prior receipt of induction chemotherapy followed by referral for concurrent chemoradiation is allowed
* Adequate lung function indicated by forced expiratory volume at 1 second (FEV1) >= 1 L is required
* The primary tumor and/or regional lymph nodes must be evaluable radiographically
* The gross target volume (GTV) is suitable for motion management using 4 dimensional computed tomography (4D CT), internal target volume (ITV), or respiratory gating; in addition, the target coverage and normal tissue constraints must be met as specified in protocol accounting for the respiratory motion of anatomy as a whole (not just the tumor)
* No prior radiation to the mediastinal structures
* Hemoglobin >= 9.0 g/dL
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Total bilirubin =< 1.5 times the upper limit of normal (ULN)
* Alanine and aspartate transaminases (ALT and AST) =< 2.5 times the ULN (=< 5 x ULN for patients with liver involvement)
* Creatinine =< 1.5 times ULN
* Patients must sign an informed consent indicating that they are aware of the investigational nature of the study in keeping with the policy of MD Anderson Cancer Center (MDACC)

Exclusion Criteria:

* Prior radiotherapy to any anatomic regions that would result in overlap of radiation dose distribution to critical structures (esophagus, heart, spinal cord, brachial plexus)
* T4 tumor with direct invasion of esophagus, spinal cord, major blood vessel, or heart
* Pregnancy
* Patients of childbearing potential must practice appropriate contraception
* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2012-09-17 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) for intensity-modulated photon therapy (IMRT) (Phase I) | 90 days
  Will be defined as the highest simultaneous integrated boost volume (SIBV) dose that has posterior probability of dose-limiting toxicity (DLT) =< 30%. DLT are defined as Common Terminology Criteria for Adverse Events (CTCAE) 4.0 grade 3+ acute radiation toxicity, including esophagitis, pneumonitis, and skin reaction that are definitely, or probably related to radiation treatment. Toxicities will be tabulated by dose, severity, and relationship to radiation therapy.
MTD for intensity-modulated proton therapy (IMPT) (Phase I) | 90 days
  Will be defined as the highest SIBV dose that has posterior probability of DLT =< 30%. DLT are defined as CTCAE 4.0 grade 3+ acute radiation toxicity, including esophagitis, pneumonitis, and skin reaction that are definitely, or probably related to radiation treatment. Toxicities will be tabulated by dose, severity, and relationship to radiation therapy.
Survival free of grade >= 3 toxicity (with a target of at least 75%) (Phase II) | 6 months
Local progression-free survival (75% at 6 months) d (Phase II) | 6 months
  Will be defined as tumor recurrence or progression inside or at the boundary of the volume defined by the 60 Gy (relative biological effectiveness) isodose line. A Bayesian method will be applied.

SECONDARY OUTCOMES:
Time to local failure (Phase II) | Up to 5 years
  The product-limit estimator of Kaplan and Meier will be used.
Progression-free survival (Phase II) | Up to 5 years
  The product-limit estimator of Kaplan and Meier will be used.
Overall survival (Phase II) | Up to 5 years
  The product-limit estimator of Kaplan and Meier will be used.
Posterior probability that the DLT rate 90 days from day 1 of radiation therapy is more than 30% (Phase II) | 90 days
  A 90% credible interval will be reported for this rate. Toxicities will be tabulated by severity and relationship to radiation therapy.
Changes in selected biomarkers (Phase II) | Baseline to up to 5 years
  Correlate changes in peripheral blood biomarkers (genes, ctDNA, microRNA, exosomes, proteins) and the study endpoints. Cox proportional hazards regression will be used to estimate the relationship between changes in selected biomarkers and time to local failure, progression-free survival, and overall survival.
Change in symptom burden using European Quality of Life Five Dimension [EQ-5D]) (Phase II) Survey | Up to 10 minutes
  Descriptive statistics and box plots will be used and will be measured by participants answers to the survey.
Change in symptom burden using MD Anderson Symptom Inventory [MDASI]-Plus Survey | Up to 10 minutes
  Descriptive statistics and box plots will be used and will be measured by participants answers to the survey.

CONTACTS AND LOCATIONS:
Overall Officials: Zhongxing Liao, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org